CLINICAL TRIAL: NCT05025631
Title: A Phase II Study on Dose Optimization of Fruquintinib in Elderly Metastatic Colorectal Cancer Patients Refractory to Standard Treatment
Brief Title: A Phase II Study on Dose Optimization of Fruquintinib in Elderly mCRC Patients Refractory to Standard Treatment（DOFEMCRC）
Acronym: DOFEMCRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhen-Yu Ding (Other)
Responsible Party: Sponsor-Investigator, Zhen-Yu Ding, Professor, Sichuan University
Organization: Sichuan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C110
Record Dates: First submitted 2021-08-25; First posted 2021-08-27 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib dose-optimization (Experimental): Fruquintinib was administered orally on 21 consecutive days in a 28-day treatment cycle. All patients were dose-optimized for the first cycle of fruquintinib - oral fruquintinib 3 mg/day in the first week; if tolerated, oral fruquintinib 4 mg/day in the second week; if still tolerated, then the dose was increased to 5 mg/day in the third week. From the second cycle, patients were given the maximum dose that they have tolerated in the first cycle.
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib was administered for 21 consecutive days of a 28-day treatment cycle. The starting dose of fruquintinib was 3 mg/day, weekly incremental dose escalation occurred up to the maximum of 5 mg/day if no significant drug-related toxicities were observed. The highest tolerated dose from cycle 1 would be administered in cycle 2 and all subsequent cycles.

SUMMARY:
A Phase II study on dose optimization of fruquintinib in elderly metastatic colorectal cancer patients refractory to standard treatment.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single arm, phase II study. In this study, the low-dose initial dose incremental optimization scheme was used in the first cycle in patients ≥65 years old who need to receive fruquintinib. The aim is to observe the safety, tolerability and efficacy of fruquintinib in elderly patients with mCRC refractory to standard treatment. The correlation between the efficacy, toxicity and geriatric evaluation of fruquintinib will also be analysed.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years and older;
2. Histologically or cytologically confirmed unresectable metastatic colorectal cancer refractory to or unfit for standard therapies;
3. ECOG PS 0-1;
4. At least 4 weeks after the last anti-tumor therapy (chemotherapy, radiotherapy, biotherapy or hormone therapy) and more than 3 months after operation treatment before enrollment;
5. Life expectancy ≥ 3 months;
6. Cooperative in observation of adverse events and curative effect;
7. No other anti-tumor concomitant treatment (including steroid drugs);
8. Adequate organ and bone marrow functions;
9. At least one measurable lesion(s);
10. Signed the written informed consent and completed the geriatric questionnaire (G8 screening form) at the time of enrollment.

Exclusion Criteria:

1. Active upper gastrointestinal ulcer, obvious vomiting, chronic diarrhea, intestinal obstruction, absorption disorder, etc which may affect drug absorption, distribution, metabolism, or clearance;
2. Evidence of central nervous system metastasis;
3. One of the following complications: uncontrolled hypertension, coronary artery disease, arrhythmia and heart failure;
4. Abuse of alcohol or drugs;
5. Less than 4 weeks from the last clinical trial;
6. Previous treatment with VEGFR inhibitors;
7. Severe uncontrolled disability with concurrent infection;
8. Proteinuria ≥ 2 + (1.0g / 24hr);
9. Uncontrollable gastrointestinal bleeding;
10. Arterial / venous thromboembolic events such as cerebrovascular accident (including transient ischemic attack) occurred within 12 months before the first dose;
11. Acute myocardial infarction, acute coronary syndrome or coronary artery bypass grafting occurred within 6 months before the first dose;
12. Fracture or wound that has not been cured for a long time;
13. Coagulation dysfunction, bleeding tendency or receiving anticoagulation treatment;
14. Congenital or acquired immune deficiency (such as HIV infection), or active hepatitis (HBV DNA ≥ 103copies / ml after regular antiviral therapy);
15. Patients who are not suitable for the study judged by the researchers.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
PFS | about a year
  Progression-free survival is determined from the date of treatment to PD or death from any cause

SECONDARY OUTCOMES:
Safety and tolerability | about a year
  Version 5.0 and AEs leading to dose interruption or discontinuation.
ORR | about a year
  Objective Response Rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version. 1.1
DCR | about a year
  Disease Control Rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version. 1.1
OS | about a year
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up
Correlation between geriatric assessment and efficacy and safety | about a year
  Statistical results obtained by analyzing the patient's geriatric assessment against efficacy and safety

CONTACTS AND LOCATIONS:
Locations (1):
- China West Hospital, Chengdu, Sichuan, China